CLINICAL TRIAL: NCT05177406
Title: Healthcare Costs and Resource Utilization in Aimovig Migraine Patients: a Retrospective Study Using United States Claims Data
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAMG334A2029
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Migraine
Keywords: Migraine,; Erenumab,; Aimovig
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Full cohort: patients newly initiating Aimovig therapy
  Interventions: Other: Aimovig

INTERVENTIONS:
Other: Aimovig — patients newly initiating Aimovig therapy
  Other Names: Erenumab

SUMMARY:
The proposed study is a retrospective, non-interventional analysis that uses medical and pharmacy claims data in the US from Komodo Health

DETAILED DESCRIPTION:
The proposed study is a retrospective, non-interventional analysis that uses medical and pharmacy claims data in the US from Komodo Health.

Study data included adjudicated and paid medical and pharmacy claims in the US between November 1, 2017 and September 1, 2019 provided by Komodo Health.

ELIGIBILITY:
Inclusion Criteria:

General Cohort

* Adult (18 years or older)
* Newly initiating on Aimovig (no other claims during a 180-day wash-in period)
* Had continuous medical and pharmacy benefit eligibility from 180 days pre-index of Aimovig through 180-days post-index

Primary & Secondary Objectives Sub-Cohort

- Had 3 consecutive months with a claim for Aimovig (≤15 days gap between days supply and the subsequent claim to be considered consecutive)

Primary & Secondary Objectives Cost Sensitivity Analyses Sub-Cohorts

* Had continuous medical and pharmacy benefit eligibility from 180 days pre-index of Aimovig through 270-days post-index to permit assessment of cost outcomes (all-cause and migraine-related) during days 91-270 post-index
* Had continuous medical and pharmacy benefit eligibility from 180 days pre-index of Aimovig to the maximum follow-up time post-index with continuous medical and prescription insurance eligibility until the data end date (September 1, 2019)

Exclusion Criteria:

* Patients with any claim for another CGRP-targeted medication (Ajovy or Emgality) during entire study period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included the Aimovig migraine patients
Sampling Method: Non-Probability Sample
Enrollment: 1839 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in migraine-related medical and prescription costs | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  Migraine-related costs included: acute and preventive migraine-related prescription costs & drug administration costs, as well as hospitalizations, emergency room (ER) visits, outpatient visits (including urgent care), provider-office visits, and diagnostic imaging with a primary diagnosis of migraine

SECONDARY OUTCOMES:
Change in all-cause costs | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with all-cause hospitalizations or ER visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with migraine-related hospitalizations or ER visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with all-cause outpatient visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with migraine-related outpatient visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with all-cause provider-office visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with migraine-related provider-office visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with all-cause neurologist office visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with migraine-related neurologist visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with all-cause pain specialist office visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with migraine-related pain specialist office visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with all-cause physical therapy visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with migraine-related physical therapy visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with all-cause psychiatrist/psychologist visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with anxiety-related psychiatrist/psychologist visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with depression-related psychiatrist/psychologist visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with any 30-day adjusted prescription for other preventive migraine medications | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in percentage of patients with any prescriptions for acute migraine medications | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of all-cause hospitalizations or ER visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of migraine-related hospitalizations or ER visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of all-cause outpatient visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of migraine-related outpatient visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of all-cause provider-office visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of migraine-related provider-office visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of all-cause neurologist office visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of migraine-related neurologist visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of all-cause pain specialist office visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of migraine-related pain specialist office visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of all-cause physical therapy visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of migraine-related physical therapy visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of all-cause psychiatrist/psychologist visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of anxiety-related psychiatrist/psychologist visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in number of depression-related psychiatrist/psychologist visits | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in the number of 30-day adjusted prescriptions for other preventive migraine medications | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  Other preventive migraine medications included anticonvulsants, antidepressants, Botox, beta blockers, calcium channel blockers, renin-angiotensin system antagonists. The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy
Change in the number of prescriptions for acute migraine medications | From 180 days pre-index date to 180 days post-index date where index date was defined as first claim for Aimovig between 05/01/18 - 03/01/19
  Acute migraine medications included ergots, prescription NSAIDs, opioids, and triptans. The outcome was evaluated during the 180-day post-index treatment period compared to the 180-day pre-index treatment period in patients newly initiating Aimovig therapy

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States